CLINICAL TRIAL: NCT05759221
Title: A Pilot Study of Peripheral Airway Biopsy for the Diagnosis of Sarcoidosis
Brief Title: Peripheral Airway Biopsy in Sarcoidosis
Acronym: Sopranos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5279
Record Dates: First submitted 2023-02-06; First posted 2023-03-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: Sarcoidosis; Bronchoscopy
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peripheral airway biopsy arm (Experimental): All patients with clinical and radiological suspicion of sarcoidosis will be submitted to biopsy of peripheral airways (> 6th branching generation).
  Interventions: Procedure: Bronchoscopy with airway biopsy

INTERVENTIONS:
Procedure: Bronchoscopy with airway biopsy — Forceps biopsy of peripheral airways under direct endoscopic visualisation.

SUMMARY:
Airway involvement in sarcoidosis was demonstrated in a meaningful, albeit variable, proportion of patients through biopsy of the central, endoscopically visible airways. Ideally, biopsy of peripheral airways, nowadays possible with the introduction in the market of ultrathin bronchoscopes, might be associated with an increased diagnostic yield for the detection of granulomas.

DETAILED DESCRIPTION:
Sarcoidosis is a systemic disorder of unknown cause that primarily involves the lung and lymphatic systems and that is more reliably diagnosed if a compatible clinical picture is combined with a pathologic demonstration of non-necrotizing epithelioid-cell granulomas. Endobronchial biopsy (EBB), taken from the central airways with standard-sized videobronchoscopes, has long been used in clinical practice, although its diagnostic yield has been shown to be widely variable across different ethnicities. A recent prospective study shows that the diagnostic yield of EBB in a sarcoidosis population with large prevalence of white Europeans is 37% overall, and 22% in patients who do not have endobronchial abnormalities. The diagnostic yield of biopsies taken from peripheral airways with ultrathin bronchoscopes was never been evaluated, to our knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Necessity of a pathological confirmation of the clinical and radiological (CT) diagnosis of sarcoidosis.
* Age >18 years
* American Society of Anesthesiologists score 1-3.

Exclusion Criteria:

* Inability of unwillingness to consent
* Steroid therapy (at least 1 week) in the 2 months preceding bronchoscopy.
* Pregnancy.
* Uncontrolled coagulopathy
* Contraindication to the temporary interruption of anticoagulants or antiplatelet drugs, except aspirin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of peripheral airway biopsy for the detection of granulomas | 1 month
  The diagnostic yield will be calculated on a per patient basis (number of patients in whom the pathological examination of peripheral airway biopsy shows non necrotizing granulomas/all the patients submitted to the sampling procedure).

SECONDARY OUTCOMES:
Complication rate | 1 day
  Incidence of early complications
Diagnostic yield for the detection of endobronchial granulomas according to sex | 6 months
  The association between the sex (male vs female) and the diagnostic yield of peripheral airway biopsy will be assessed
Diagnostic yield for the detection of endobronchial granulomas according to the ethnicity | 6 months
  The association between the ethnicity (white versus other) and the diagnostic yield of peripheral airway biopsy will be assessed
Diagnostic yield for the detection of endobronchial granulomas according to the history of malignancy | 6 months
  The association between a history of malignancy (presence versus absence of any malignancy diagnosed within 5 years of the procedure) and the diagnostic yield of peripheral airway biopsy will be assessed
Diagnostic yield for the detection of endobronchial granulomas according to the sarcoidosis stage | 6 months
  The association between the sarcoidosis stage at CT (I vs II vs II vs IV) and the diagnostic yield of peripheral airway biopsy will be assessed
Diagnostic yield for the detection of endobronchial granulomas according to the presence of large airway mucosal abnormalities | 6 months
  The association between the presence of endoscopically visible large airway abnormalities and the diagnostic yield of peripheral airway biopsy will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Univeristario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No